CLINICAL TRIAL: NCT04398186
Title: The Effect of Polycystic Ovary Syndrome on Pelvic Floor Structure and Function
Status: Completed | Type: Observational
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, Sebnem Alanya Tosun, Assistant Professor, Giresun University
Other Study IDs: GiresunU
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Reproductive System Disorder; Urinary Incontinence; Urogenital Disease; Polycystic Ovary Syndrome
Keywords: polycystic ovary syndrome; urinary incontinence; anogenital distance
MeSH Terms: conditions — Urinary Incontinence; Urogenital Diseases; Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Study group 1: Hiperandrogenism + ultrasonographic PCO
  Interventions: Diagnostic Test: Anogenital distance measurement
- Study group 2: Menstruel cycle irregular + ultrasonographic PCO
  Interventions: Diagnostic Test: Anogenital distance measurement
- Study group 3: Menstruel cycle irregular + ultrasonographic PCO + hyperandrogenism
  Interventions: Diagnostic Test: Anogenital distance measurement
- Control group: Do not have PCOS
  Interventions: Diagnostic Test: Anogenital distance measurement

INTERVENTIONS:
Diagnostic Test: Anogenital distance measurement — Measurements of AGD and perineal muscle strength

SUMMARY:
Polycystic Ovarian Syndrome (PCOS) is the most common endocrinological disorder in women of reproductive age, and its prevalence is reported to be 6-21% in women aged 15-49 (1). Although its etiopathogenesis is still not clear, it is known that it is due to the disregulation of ovarian steroidogenesis under the influence of some environmental and genetic factors. Diagnosis of ESHRE / ASRM has set Rotterdam criteria in 2003; one of these criteria is the presence of hyperandrogenism (2). Hyperandrogenism leads to an increase in general muscle mass in the body (1, 3, 4).

Pelvic floor muscles are associated with urethra in the anterior compartment, rectum and anus in the posterior compartment, and uterine support in the apex; major urinary and fecal continence ensuring its functions in order to stop in the appropriate position of the pelvic organs (5). The well-being of the pelvic floor muscle strength has a protective effect from urinary and fecal incontinence.

It has been emphasized that the "anogenital distance" determined by the measurement of the anal region anterior to the clitoris anterior may also be a criteria in the diagnosis of Polycystic Ovary Syndrome (7,8,9).

In this study, patients in the reproductive age between 18-40 years, who applied to our gynecology outpatient clinic and were diagnosed as PCOS according to Rotterdam criteria wil be study gorup and the women without PCOS will be control group. We aimed to evaluate the pelvic muscle strength with perineometry, to measure anogenital distance and to determine possible relationships with each other. In addition to demographic information, ICIQ-SF (Urinary incontinence inquiry short form) will also be taken to evaluate pelvic floor function (10).

ELIGIBILITY:
Inclusion Criteria:

* Nulliparity

Exclusion Criteria:

* Endocrine disorders
* Anabolic drug usage Multiparity

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Reproductive aged females
Study Population: Reproductive aged females, age between 18-40 yrs.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Anogenital distance measurement in PCOS | 01.06.2020- 01.11.2020

CONTACTS AND LOCATIONS:
Locations (1):
- Sebnem Alanya Tosun, Giresun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided